CLINICAL TRIAL: NCT02697721
Title: Optimization of "Powerful Tools for Caregivers" of Dementia Patients
Brief Title: Powerful Tools for Caregivers of Dementia Patients
Acronym: PTC-dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Antonio Terracciano, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6AZ09
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Caregivers; Dementia; Alzheimer Disease
Keywords: Caregivers; Behavioral symptoms; Dementia; Alzheimer disease; Physical activity; Depressive symptoms; Powerful Tools for Caregivers; Chronic Disease Self-Management Program
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavioral Symptoms; Motor Activity; Depression | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Powerful Tools for Caregivers (Experimental): A 6-week psycho-educational program
  Interventions: Behavioral: Powerful Tools for Caregivers
- Control group, delayed intervention (Other): Control group with delayed intervention
  Interventions: Other: Control with delayed intervention

INTERVENTIONS:
Behavioral: Powerful Tools for Caregivers — Powerful Tools for Caregivers is a 6-week psychoeducational program. Each week the caregivers will attend a 90-minute workshop in a group setting. These sessions will be co-led by two trained and certified leaders who follow the scripted program. In addition to providing education about caregiving and the importance of self-care, the classes will help caregivers develop self-care tools to manage personal stress and improve communication skills.
  Arms: Powerful Tools for Caregivers
Other: Control with delayed intervention — Control with delayed intervention
  Arms: Control group, delayed intervention

SUMMARY:
The purpose of this study is to examine if a psycho-educational intervention for caregivers of patients with dementia will decrease caregiver burden, increase caregiver physical activity, and decrease the reporting of behavioral and psychological symptoms of the person with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver lives with or provides care for the care recipient for an average of at least 4 hours per day.
* Care for an individual with a physician diagnosis of dementia (mild to moderate stage of dementia).
* Care for a care recipient who experiences behavioral symptoms that bother or upset the caregiver moderately, very much, or extremely. The occurrence of problematic behaviors and caregivers' reactions will be assessed with 6-items adapted from the Revised Memory and Behavior Problems Checklist (Teri et al 1992).

Exclusion Criteria:

* Care for a care recipient who is bed-bound or has advanced dementia: Functional Assessment Staging (FAST)(Sclan & Reisberg 1992) stage 7.
* Caregiver's cognitive, hearing, visual, or other physical impairments lead to difficulty with informed consent process, assessment, or participation in the intervention.
* Caregiver who is involved in another trial that addresses caregiver burden or behavioral expressions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden | 6 weeks
  Zarit Caregiver Burden Scale scores
Frequency and reaction to care recipient behavioral and psychological symptoms of dementia | 6 weeks
  Revised Memory and Behavior Problems Checklist scores
Frequency of care recipient agitated behaviors | 6 weeks
  Cohen-Mansfield Agitation Inventory scores

SECONDARY OUTCOMES:
Activity parameters as assessed by FitBit | 6 weeks
Depressive symptoms | 6 weeks
  Center for Epidemiologic Studies Depression Scale scores
Caregiving Self-Efficacy | 6 weeks
  Caregiving Self-Efficacy Scale scores
Self-rated health | 6 weeks
  Single item "In general, would you say your health is...." with response options from 1= poor to 5=excellent.
Life satisfaction | 6 weeks
  Single item "I am satisfied with my life" with response options from 0=Strongly disagree to 4=Strongly agree
Perceived change | 6 weeks
  Perceived Change Index score
Neuropsychiatric symptoms in care recipients | 6 weeks
  Neuropsychiatric Inventory score

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University College of Medicine, Tallahassee, Florida, United States

REFERENCES:
- [Result] Terracciano A, Artese A, Yeh J, Edgerton L, Granville L, Aschwanden D, Luchetti M, Glueckauf RL, Stephan Y, Sutin AR, Katz P. Effectiveness of Powerful Tools for Caregivers on Caregiver Burden and on Care Recipient Behavioral and Psychological Symptoms of Dementia: A Randomized Controlled Trial. J Am Med Dir Assoc. 2020 Aug;21(8):1121-1127.e1. doi: 10.1016/j.jamda.2019.11.011. Epub 2019 Dec 19. PMID 31866419